CLINICAL TRIAL: NCT01491633
Title: Phase II Trial of Dasatinib in Advanced (Stage IIIB/IV) Squamous Cell Lung Cancer
Brief Title: Dasatinib in Advanced Squamous Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety issues/concerns per DF/HCC PI
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Bruce Johnson, MD, Professor of Medicine, Harvard Medical School, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-142
Record Dates: First submitted 2011-10-05; First posted 2011-12-14 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Lung cancer; NSCLC; Stage IIIB; Stage IV
MeSH Terms: conditions — Lung Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): Dasatinib 140 mg by mouth each day
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 140 mg orally, daily in 28 day cycles
  Other Names: BMS-354825

SUMMARY:
Dasatinib is a drug that has been shown to stop some cancer cells from growing. This drug has been used in treatment for other types of cancer and information from other research studies suggests that dasatinib may help to stop squamous cell lung cancer from growing, especially in individuals whose tumor has a mutation in the DDR2 gene.

Advanced squamous cell lung cancer (SqCC) carries a poor prognosis and new therapeutic targets are needed. Several studies have examined dasatinib in NSCLC; these report significant toxicities, but also responses in patients found to harbor mutations in DDR2 or BRAF.

An open-label phase II trial with dasatinib was carried out to determine the response rates in patients with SqCC who had previously failed standard chemotherapy and to correlate responses with patient genotype.

DETAILED DESCRIPTION:
Dasatinib will be taken orally, daily in cycles of 28 days.

On the first day of study treatment and at 2 weeks, 4 weeks and then every 4 weeks subjects will have the following:

* Medical history and clinical exam
* Safety blood tests
* Measurement of Performance Status
* Review of pill log
* CT scans will be done every 8 weeks.

In this research study, the investigators are looking at how well dasatinib works in treating squamous cell lung cancer.

Dasatinib administered at 140mg per day for the treatment of advanced SqCC of the lung is associated with excess adverse events, similar to other studies, so is not recommended in unselected patients. Further work to identify patients likely to benefit from dasatinib and in managing dasatinib-related toxicities is needed.

ELIGIBILITY:
Inclusion Criteria:

* Stage III/B or IV squamous NSCLC
* Measurable disease
* Previously offered all standard chemotherapy regimens for advanced squamous cell lung cancer
* ECOG performance status of 0 or 1
* Estimated life expectancy greater than 12 weeks
* Normal organ and marrow function
* Confirmed availability of archival pathology samples
* Agrees to discontinue St. Johns Wort
* Able to take medications by mouth
* Willing and able to use acceptable method of birth control for the entire study period and for at least 4 weeks after the last dose of study drug

Exclusion Criteria:

* Pregnant or breast-feeding
* Chemotherapy or radiotherapy within 4 weeks prior to entering study
* Receiving any other investigational agents
* Known untreated or progressive brain metastases
* History of prior treatment with or allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib, nilotinib or imatinib
* Taking medications known to be potent CYP3A4 inhibitors
* Currently taking H2 inhibitors or proton pump inhibitors
* Currently taking drugs or have taken drugs in the past 7 days that are generally accepted to have a risk of causing Torsades de Pointes
* HIV positive
* Clinically uncontrolled hypertension (blood pressure > 160/110)
* Previous or concurrent malignancy except adequately treated basal or squamous cell skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 5 years
* Active and uncontrolled clinically significant infection
* Chronic gastrointestinal disease
* Acquired or congenital bleeding disorder or clinically significant gastrointestinal bleeding within 3 months
* Supplemental oxygen required for current malignancy
* Evidence of symptomatic pleural effusions unless undergoing a therapeutic thoracentesis as part of non-study care
* Individuals who are prisoners or who are compulsory detained for medical or psychiatric reasons
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Hypokalemia or hypomagnesemia that cannot be corrected prior to dasatinib administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Johnson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Brunner AM, Costa DB, Heist RS, Garcia E, Lindeman NI, Sholl LM, Oxnard GR, Johnson BE, Hammerman PS. Treatment-related toxicities in a phase II trial of dasatinib in patients with squamous cell carcinoma of the lung. J Thorac Oncol. 2013 Nov;8(11):1434-7. doi: 10.1097/JTO.0b013e3182a47162. PMID 24128713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dasatinib
Started | 5
Completed | 0
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 59 [55 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Determine the overall response rate of patients with squamous cell carcinoma of the lung treated with dasatinib
Time Frame: 2 years
Measure: Number; unit: percent
Arm/Group | Dasatinib
Number analyzed (Participants) | 5
percent | NA — No subjects were evaluable for response

2. Secondary Outcome: Types and Frequency of DDR2 Mutations
Description: Determine frequency of DDR2 mutations in study patients
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 5
participants | 0

3. Secondary Outcome: Survival
Description: Establish the overall survival of patients with SCC treated with dasatinib
Time Frame: 2 years
Population: One subject who was alive at the end of the study was censored from the survival analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dasatinib
Number analyzed (Participants) | 4
days | 112 (85)

4. Secondary Outcome: Toxicities
Description: Define the toxicities of dasatinib when administered to the patient population. NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 will be utilized for adverse event reporting.
Time Frame: 2 years
Measure: Number; unit: grade 3 toxicities
Arm/Group | Dasatinib
Number analyzed (Participants) | 5
grade 3 toxicities | 3

5. Post Hoc Outcome: Time on Study
Description: Number of days participant remained on study
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dasatinib
Number analyzed (Participants) | 5
days | 22 (12)

ADVERSE EVENTS:
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=5)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Elevated LFTs (Gastrointestinal disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the toxicity of the study agent no subjects were evaluable for response

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No